CLINICAL TRIAL: NCT03721094
Title: Cognitive Load and Performance in Immersive Virtual Reality Versus Conventional Virtual Reality Simulation Training of Laparoscopic Surgery - a Randomized Trial
Brief Title: Training Using Immersive Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Joakim Grant Frederiksen, Principal Investigator, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HMD-VR
Record Dates: First submitted 2018-10-05; First posted 2018-10-26 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Cognitive Load, Performance

STUDY DESIGN:
Intervention Model Description: A single-center randomized trial was designed according to the CONSORT statement
Masking Description: Participants and the principal investigators were blinded to performance metrics by the simulator during the supervised procedure and the three test procedures. Participants and the data collector could not be blinded to the allocation/intervention. The investigator in charge of the statistical analysis was blinded to participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive virtual reality (Other): Completing the procedures in immersive virtual reality
  Interventions: Other: Immersive virtual reality
- Conventional virtual reality (No Intervention): Completing the procedures in conventional virtual reality

INTERVENTIONS:
Other: Immersive virtual reality — In the IVR environment, four different 360-degrees videos were in sequence played as backdrop during the procedure. The videos reflected real life situations in the operating room with two videos representing calm periods, one video representing a light stressor and one video representing a severe stressor with a bleeding (2 ml/s) being triggered in the simulation. Participants complete the procedures while wearing the head mounted device.
  Arms: Immersive virtual reality

SUMMARY:
In this study, the investigators examine the cognitive load (CL) and performance of a laparoscopic procedure in immersive virtual reality and controlled virtual reality in a randomized, controlled setup. Virtual reality (VR) simulators combined with head mounted displays (HMDs) enable highly immersive virtual reality (IVR) for surgical skills training, potentially bridging the gap between the simulation environment and real-life operating room (OR) conditions. However, the increased complexity of the learning situation in IVR could potentially induce high CL thereby inhibiting performance and learning.

ELIGIBILITY:
Inclusion Criteria:

* First year resident

Exclusion Criteria:

* Previous participation in trials involving laparoscopic training
* Prior experience with laparoscopic surgery (having performed one or more laparoscopic procedures as primary surgeon, including supervised procedures)
* Not speaking Danish on a conversational level

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Cognitive load | 6 months
  Measurement of the participants cognitive load during four different time periods during the three procedures. Cognitive load was estimated by secondary-task reaction time. The investigators used an external and commercially available reaction timer (American Educational Products LLC, USA) to measure participants response time (in hundreds seconds) to an auditory stimulus (a beep). Reaction time was measured before and after the simulation to provide an individual baseline, and during the simulation at t=80 s, t=130 s, t=180 s and t=240 s. All reaction time measurements were done in series of four repeated measurements. It was also noted if the reaction time was measured while the participant was using the foot pedal for cauterization in the simulation.

SECONDARY OUTCOMES:
Time to completion of procedure | 6 months
  Time to completion of procedure (measured in seconds)
Diathermy damage | 6 months
  Damage to surrounding tissue during the procedure (in number of incidents)
Blood loss | 6 months
  Blood loss during the procedure (in ml)
Efficience of instrument movements (length) | 6 months
  Measurement of movement of the left and right hand in meters
Efficience of instrument movements (degrees) | 6 months
  Measurement of angular movements of the left and right hand in degrees

OTHER OUTCOMES:
Motion sickness | 6 months
  Motion sickness was assessed using a post-procedure questionnaire. The investigators used the MSAQ (Motion Sickness Assesment Questionnaire) developed by Gianaros et al in 2001. The questionnaire consisted of 16 statements and the participants had to rate how accurately the statements describe their experience in a numbered scale from 1 (not at all) to 9 (severely). The 16 statements were divided into for categories: Gastrointestinal; Central; Peripheral; Sopite-related. The overall motion sickness score was obtained by calculating the percentage of total points scored: (sum of points from all items/144) * 100. Subscale scores was obtained by calculating the percent of points scored within each factor: (sum of gastrointestinal items/36) * 100; (sum of central items/45) * 100; (sum of peripheral items/27) * 100; (sum of sopite-related items/36) * 100.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Konge, PhD, Study Director — Copenhagen Academy for Medical Education and Simulation
Locations (1):
- Copenhagen Academy for Medical Education and Simulation, Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sorensen SM, Savran MM, Konge L, Bjerrum F. Three-dimensional versus two-dimensional vision in laparoscopy: a systematic review. Surg Endosc. 2016 Jan;30(1):11-23. doi: 10.1007/s00464-015-4189-7. Epub 2015 Apr 4. PMID 25840896
- [Background] Nagendran M, Gurusamy KS, Aggarwal R, Loizidou M, Davidson BR. Virtual reality training for surgical trainees in laparoscopic surgery. Cochrane Database Syst Rev. 2013 Aug 27;2013(8):CD006575. doi: 10.1002/14651858.CD006575.pub3. PMID 23980026
- [Background] Moorthy K, Munz Y, Adams S, Pandey V, Darzi A. A human factors analysis of technical and team skills among surgical trainees during procedural simulations in a simulated operating theatre. Ann Surg. 2005 Nov;242(5):631-9. doi: 10.1097/01.sla.0000186298.79308.a8. PMID 16244534
- [Background] van Merrienboer JJ, Sweller J. Cognitive load theory in health professional education: design principles and strategies. Med Educ. 2010 Jan;44(1):85-93. doi: 10.1111/j.1365-2923.2009.03498.x. PMID 20078759
- [Background] Huber T, Paschold M, Hansen C, Wunderling T, Lang H, Kneist W. New dimensions in surgical training: immersive virtual reality laparoscopic simulation exhilarates surgical staff. Surg Endosc. 2017 Nov;31(11):4472-4477. doi: 10.1007/s00464-017-5500-6. Epub 2017 Apr 4. PMID 28378077
- [Background] Andersen SA, Mikkelsen PT, Konge L, Caye-Thomasen P, Sorensen MS. Cognitive Load in Mastoidectomy Skills Training: Virtual Reality Simulation and Traditional Dissection Compared. J Surg Educ. 2016 Jan-Feb;73(1):45-50. doi: 10.1016/j.jsurg.2015.09.010. Epub 2015 Oct 21. PMID 26481267
- [Background] Strandbygaard J, Bjerrum F, Maagaard M, Winkel P, Larsen CR, Ringsted C, Gluud C, Grantcharov T, Ottesen B, Sorensen JL. Instructor feedback versus no instructor feedback on performance in a laparoscopic virtual reality simulator: a randomized trial. Ann Surg. 2013 May;257(5):839-44. doi: 10.1097/SLA.0b013e31827eee6e. PMID 23295321
- [Background] Thorson CM, Kelly JP, Forse RA, Turaga KK. Can we continue to ignore gender differences in performance on simulation trainers? J Laparoendosc Adv Surg Tech A. 2011 May;21(4):329-33. doi: 10.1089/lap.2010.0368. PMID 21563940
- [Background] White MT, Welch K. Does gender predict performance of novices undergoing Fundamentals of Laparoscopic Surgery (FLS) training? Am J Surg. 2012 Mar;203(3):397-400; discussion 400. doi: 10.1016/j.amjsurg.2011.09.020. PMID 22364906
- [Background] Gianaros PJ, Muth ER, Mordkoff JT, Levine ME, Stern RM. A questionnaire for the assessment of the multiple dimensions of motion sickness. Aviat Space Environ Med. 2001 Feb;72(2):115-9. PMID 11211039

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT03721094/Prot_SAP_000.pdf